CLINICAL TRIAL: NCT03995810
Title: Oral Carnosine for Neuromuscular Performance, Brain Biomarkers of Carnosine Metabolism and Health-related Quality of Life in Multiple Sclerosis
Brief Title: Oral Carnosine for Neuromuscular Performance in Multiple Sclerosis
Acronym: CARMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Collaborators: CarnoMed (Unknown)
Responsible Party: Principal Investigator, Sergej Ostojic, University Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CM-03CS/2019
Record Dates: First submitted 2019-06-18; First posted 2019-06-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Carnosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carnosine (Experimental): Carnosine, capsulle, 2 g/day, 8 weeks
  Interventions: Dietary Supplement: Carnosine, capsulle, 2 g/day, 8 weeks

INTERVENTIONS:
Dietary Supplement: Carnosine, capsulle, 2 g/day, 8 weeks — We will administer supplemental carnosine (2 grams per day) for 8 weeks

SUMMARY:
Low levels of tissue carnosine and mitochondrial dysfunction appears to accompany multiple sclerosis (MS), with oral carnosine might be applicable to tackle impaired bioenergetics and oxidative stress in MS, and perhaps win back neuromuscular function. However, several formulations of carnosine have shown limited applicability due to restraints in brain delivery or tissue performance. No human studies so far evaluated the impact of innovative carnosine formulation (Karnozin EXTRA) in MS. Here, we will evaluate the impact of supplemental carnosine on neuromuscular performance, brain biomarkers of carnosine metabolism, and health-related quality of life in a case series of patients with MS.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a complex autoimmune disorder that affects millions of people around the world, negatively interfering with different aspects of health and everyday life. Being the most frequently seen demyelinating disease, MS prevalence varies considerably, from high levels in North America and Europe (> 100/100,000 inhabitants) to low rates in Eastern Asia and sub-Saharan Africa (2/100,000 population). Due to its rather high prevalence in developed countries, the development of effective and applicable strategies to prevent or manage MS becomes a must for the medical community. Among other factors, it appears that low levels of tissue carnosine and mitochondrial dysfunction accompany MS, with oral carnosine might be applicable to tackle impaired bioenergetics and oxidative stress in MS, and perhaps win back neuromuscular function. However, several formulations of carnosine have shown limited applicability due to restraints in brain delivery or tissue performance thus pushing both industry and researchers to find bioavailable and effective formulation of carnosine. No human studies so far evaluated the impact of innovative carnosine formulation (Karnozin EXTRA) in MS. Here, we will evaluate the impact of supplemental carnosine on neuromuscular performance, brain biomarkers of carnosine metabolism, and health-related quality of life in a case series of patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body mass index 19 - 30 kg/m2
* Free of major chronic diseases or acute disorders besides MS
* Fulfilled 2017 McDonald Criteria for the diagnosis of MS

Exclusion Criteria:

* Pregnancy
* Psychiatric comorbidity
* Use of dietary supplements within 4 weeks before study commences
* Unwillingness to return for follow-up analysis
* Abnormal values for lab clinical chemistry (> 2 SD)
* Immunotherapy for the past 6 months
* Treated with systemic corticosteroids during the 30 days before study commences

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Brain carnosine change | Baseline vs. eight weeks
  Monitor change in brain carnosine levels

SECONDARY OUTCOMES:
Health-related quality of life with SF36 Questionnaire change | Baseline vs. eight weeks
  Monitor change in health-related quality of life with SF36 Questionnaire
Change in neuromuscular performance for autonomic dysfunction (Ewing) | Baseline vs. eight weeks
  Monitor change in neuromuscular performance for autonomic dysfunction (Ewing)
Change in multidimensional fatigue | Baseline vs. eight weeks
  Monitor change in multidimensional Multidimensional Fatigue Inventory (MFI) 20-item questionnaire
Change in blood clinical chemistry panel | Baseline vs. eight weeks
  Lactic acid change in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Principal Investigator — University of Novi Sad
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after request to PI
Supporting Information: Study Protocol
Time Frame: Six months after a completion of the study.
Access Criteria: No specific sharing access criteria

REFERENCES:
- [Background] Keytsman C, Blancquaert L, Wens I, Missine M, Noten PV, Vandenabeele F, Derave W, Eijnde BO. Muscle carnosine in experimental autoimmune encephalomyelitis and multiple sclerosis. Mult Scler Relat Disord. 2018 Apr;21:24-29. doi: 10.1016/j.msard.2018.02.013. Epub 2018 Feb 11. PMID 29454153
- [Background] Sariev AK, Abaimov DA, Tankevich MV, Pantyukhova EY, Prokhorov DI, Fedorova TN, Lopachev AV, Stvolinskii SL, Konovalova EV, Seifulla RD. [Experimental study of the basic pharmacokinetic characteristics of dipeptide carnosine and its efficiency of penetration into brain tissues]. Eksp Klin Farmakol. 2015;78(3):30-5. Russian. PMID 26036009